CLINICAL TRIAL: NCT04937920
Title: A Randomized, Double-Blinded, Aqueous Gel-Controlled Dose Escalating Trial to Study the Safety and Antimicrobial Efficacy of DBI-002 Probiotic vs. Aqueous Gel and Vehicle Gel vs. Aqueous Gel in Adults With Tinea Versicolor
Brief Title: A Trial to Evaluate the Safety and Antimicrobial Efficacy of DBI-002 Probiotic in Adults With Tinea Versicolor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DBI-202
Record Dates: First submitted 2021-06-01; First posted 2021-06-24 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-04

CONDITIONS: Tinea Versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — BANG polymer gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBI-002 probiotic gel (Active Comparator): Topical application of DBI-002 probiotic gel on skin affected with tinea versicolor
  Interventions: Biological: DBI-002 probiotic gel
- Aqueous gel (Placebo Comparator): Topical application of aqueous gel on skin affected with tinea versicolor
  Interventions: Biological: Aqueous gel

INTERVENTIONS:
Biological: DBI-002 probiotic gel — Topical application on skin affected with tinea versicolor
  Arms: DBI-002 probiotic gel
Biological: Aqueous gel — Topical application on skin affected with tinea versicolor
  Arms: Aqueous gel

SUMMARY:
A Randomized, Double-Blinded, Aqueous Gel-Controlled Dose Escalating Trial to Study the Safety and Antimicrobial Efficacy of DBI-002 Probiotic vs. Aqueous Gel and Vehicle Gel vs. Aqueous Gel in Adults with Tinea Versicolor (DBI-202).

DETAILED DESCRIPTION:
All subjects are required to have a clinical diagnosis of Tinea Versicolor on their chest and back. Each subject will serve as their own control, with aqueous gel applied to the chest or back, and the non-aqueous gel (DBI-002 or vehicle) applied to the opposite side. Treatment kits will be assigned sequentially to subjects. The subject and the investigator will be blinded to the pre-defined randomization assignments.

In this Phase IIA proof-of-mechanism study, cohorts 1, 2, and 3 were designed to be similar to a dose-escalating study. These cohorts will be enrolled sequentially, with a safety pause in between cohorts to evaluate events and/or local tolerability to topical application of the investigational product (DBI-002) or aqueous gel. Within each cohort, the first two subjects enrolled will have a single application of DBI-002 and aqueous gel, with a pause to assess adverse events and local tolerability. In the absence of safety concerns, the remaining subjects in that cohort will be enrolled to receive five consecutive daily applications of DBI-002 and aqueous gel. Cohort 1 will be low dose. Cohort 2 will be medium dose. Cohort 3 will be high dose. In the absence of safety concerns, the Investigator will proceed to enroll the next cohort, or extend (EXT) the enrollment of a cohort upon receiving Ethics Committee approval. Single-dose subjects remain in their original single-dose cohort assignment and do not dose-escalate, nor participate in the multiple-dose portion of that cohort, nor Cohort 4.

The fourth cohort, Cohort 4, was designed to compare vehicle with aqueous gel. All subjects in this cohort will be required to receive five consecutive daily applications of vehicle and aqueous gel. The Investigator may enroll cohort 4 in parallel with the above cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand, agree to and sign the study Informed Consent Form (ICF). If the subject is unable to provide consent him/herself, the subject's legally acceptable representative may provide written consent.
2. Male or Female Subjects of any race 18 - 65 years of age.
3. Subjects with a clinical diagnosis of Tinea versicolor (TV is a common benign superficial cutaneous fungal infection usually characterized by hypopigmented or hyperpigmented macules and patches on the chest and back).
4. A positive potassium hydroxide (KOH) examination consistent with Malassezia prior to the treatment period done at the clinical site.
5. Agree to not use soap and water on the chest and back for at least 12 hours before the study visits for Baseline/Day 1, Day 5, and Day 14, and follow all study instructions for use of soap and water on the chest and back during participation in the study.

Exclusion Criteria:

1. Females who are pregnant, planning a pregnancy, or breastfeeding.
2. Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the patient to an unacceptable risk by study participation.
3. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see below).
4. Known sensitivity to any of the components of the study medication.
5. Use of a prescription or non-prescription topical treatment on the targeted TV anatomical locations within the previous 4 weeks, for example: anti-fungal, antibacterial or anti-microbial products, selenium and anti-inflammatories (e.g., corticosteroids).
6. Use of a systemic anti-fungal or antibiotic treatment for TV within the previous 4 weeks, Use of medicated shampoos and/or soaps within the previous 4 weeks.
7. Treatment of any type of cancer within the last 6 months.
8. History of any significant internal disease which contraindicates use of live microbiome (e.g. leukemia, liver failure, cardiovascular disease).
9. Subjects who are known to be allergic to any of the test product(s) or any components in the investigational product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure (IB).
10. AIDS or AIDS related complex by medical history.
11. Known or suspected use of immunosuppressive medications and/or has a known or suspected autoimmune disease.
12. Any subject not able to meet the study attendance requirements.
13. Subjects who have participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Zepeda, MD, Principal Investigator — Zepeda Dermatologia
Locations (1):
- Zepeda Dermatologia, Santa Tecla, La Libertad Department, El Salvador

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects are required to have Tinea Versicolor on their chest and back, with no pre-assignment, as each subject functions as their own control. Each subject had test article (aqueous gel and active) applied, randomized, within treatment sites to 100cm2. The dose-escalating DBI-002 cohorts (1, 2, and 3) were enrolled in sequence, with a safety pause between cohorts to assess adverse events and local reactions to topical application. 34 total subjects were enrolled and received treatment.
Units Other Than Participants: Treatment sites
Groups:
- Cohort 1: Low dose 10^6 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose (first 2 subjects) OR Once-daily application for 5 consecutive days (last 4 subjects) Safety pauses between single and multi-dose subjects, and prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort.
- Cohort 2: Medium dose 10^8 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose (first 2 subjects) OR Once-daily application for 5 consecutive days (last 4 subjects) Safety pauses between single and multi-dose subjects, and prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort.
- Cohort 3: High dose 10^10 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose (first 2 subjects) OR Once-daily application for 5 consecutive days (last 4 subjects) Safety pauses between single and multi-dose subjects, and prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort.
- Cohort 1EXT: Low dose 10^6 CFUs/ml of DBI- 002 probiotic vs. aqueous gel Once-daily application for 5 consecutive days (4 subjects) Safety pause prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort.
- Cohort 2EXT: Medium dose 10^8 CFUs /ml of DBI-002 probiotic vs. aqueous gel Once-daily application for 5 consecutive days (4 subjects) Safety pause prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort.
- Cohort 3EXT: High dose 10^10 CFUs/ml of DBI- 002 probiotic vs. aqueous gel Once-daily application for 5 consecutive days (4 subjects) Safety pause prior to enrolling next cohort. No subject is dose escalated. Subjects are enrolled in only one cohort
- Cohort 4: Vehicle gel vs. aqueous (CMC) gel
  Once-daily application for 5 consecutive days
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 1EXT | Cohort 2EXT | Cohort 3EXT | Cohort 4
Started | 6; 12 Treatment sites | 6; 12 Treatment sites | 6; 12 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites
Aqueous Gel (Back or Chest) (Each subject functions as their own control. (Subject's chest or back)) | 6; 6 Treatment sites | 6; 6 Treatment sites | 6; 6 Treatment sites | 4; 4 Treatment sites | 4; 4 Treatment sites | 4; 4 Treatment sites | 4; 4 Treatment sites
DBI-002 Probiotic (Back or Chest) (Each subject functions as their own control. (Subject's chest or back)) | 6; 6 Treatment sites | 6; 6 Treatment sites | 6; 6 Treatment sites | 4; 4 Treatment sites | 4; 4 Treatment sites | 4; 4 Treatment sites | 0; 0 Treatment sites
Vehicle Gel (Back or Chest) (Each subject functions as their own control. (Subject's chest or back)) | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 4; 4 Treatment sites
Completed | 6; 12 Treatment sites | 6; 12 Treatment sites | 6; 12 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites | 4; 8 Treatment sites
Not Completed | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites | 0; 0 Treatment sites

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1; Cohort 1EXT: Low dose 10^6 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Cohort 2; Cohort 2EXT: Medium dose 10^8 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Cohort 3; Cohort 3EXT: High dose 10^10 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 1EXT | Cohort 2EXT | Cohort 3EXT | Cohort 4 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 4 | 4 | 4 | 34
Age, Categorical [Count of Participants; unit: Participants] — Age: 18 to 65 years of age, at enrollment
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 6 | 6 | 6 | 4 | 4 | 4 | 4 | 34
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (10.6) | 24.5 (1.52) | 29.0 (8.22) | 29.0 (8.29) | 47.3 (13.6) | 31.3 (13.1) | 34.8 (13.1) | 32.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 2 | 1 | 1 | 0 | 12
  Male | 6 | 2 | 2 | 2 | 3 | 3 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 6 | 4 | 4 | 4 | 4 | 34
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  El Salvador | 6 | 6 | 6 | 4 | 4 | 4 | 4 | 34
Clinical diagnosis of Tinea Versicolor on the chest and back [Count of Participants; unit: Participants] — Clinical diagnosis of Tinea Versicolor on the chest and back, by the Investigator and KOH
  Participants | 6 | 6 | 6 | 4 | 4 | 4 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Molecular Diagnostic qPCR Comparison of DBI-002 Drug Product and Malassezia (Fungal Cause of Tinea Versicolor)
Description: The primary analysis will summarize the number of subjects with more qPCR DBI-002 drug product and more improvement in qPCR Malassezia (fungal cause of tinea versicolor) between DBI-002 Drug Product (Active) and aqueous gel (Control) at Day 5 or Day 14 versus Baseline.
Time Frame: 14 days of participation
Population: The primary analysis will compare the differences at Day 5 between DBI-002 Drug Product (DP), vehicle gel, and/or aqueous gel in abundance of Malassezia based on molecular diagnostic qPCR using a 2-sided Wilcoxon sign rank test, alpha = 0.05, with a null hypothesis of median difference equal to zero.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2EXT: Medium dose 10^8 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 1EXT | Cohort 2EXT | Cohort 3EXT
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 4 | 4
Participants
  Day 5 qPCR DBI-002 Drug Product: # Subjects where Active Improves More than Aqueous Gel (Control) | 2 | 4 | 5 | 1 | 1 | 4
  Day 14 qPCR DBI-002 Drug Product: # Subjects where Active Improves More than Aqueous Gel (Control) | 0 | 1 | 4 | 0 | 0 | 2
  Day 5 qPCR Malassezia(fungal cause of TV):# Subjects where Active Improves More than Aqueous Gel | 3 | 5 | 5 | 4 | 4 | 2
  Day 14 qPCR Malassezia(fungal cause of TV):# Subjects where Active Improves More than Aqueous Gel | 3 | 3 | 4 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 1EXT vs Cohort 2EXT vs Cohort 3EXT; The analysis compared the differences at Day 5 between DBI-002 probiotic gel (active) and vehicle gel (active Cohort 4 only) in abundance of Malassezia based on molecular diagnostic qPCR using a 2-sided Wilcoxon sign rank test, alpha = 0.05, with a null hypothesis of median difference equal to zero; Test type: Other; p = 0.2, Wilcoxon (Mann-Whitney); Mean Paired Change from Baseline = -29620
Statistical Analysis 2: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 1EXT vs Cohort 2EXT vs Cohort 3EXT; The analysis compared the differences at Day 14 between DBI-002 probiotic gel (active) and vehicle gel (active Cohort 4 only) in abundance of Malassezia based on molecular diagnostic qPCR using a 2-sided Wilcoxon sign rank test, alpha = 0.05, with a null hypothesis of median difference equal to zero; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney); Mean Paired Change from Baseline = 127195
Statistical Analysis 3: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 1EXT vs Cohort 2EXT vs Cohort 3EXT; The analysis compared the differences at Day 5 between aqueous gel (control) and vehicle gel (active Cohort 4 only) in abundance of Malassezia based on molecular diagnostic qPCR using a 2-sided Wilcoxon sign rank test, alpha = 0.05, with a null hypothesis of median difference equal to zero; Test type: Other; p = 0.6, Wilcoxon (Mann-Whitney); Mean Paired Change from Baseline = -41659
Statistical Analysis 4: Comparison: Cohort 1 vs Cohort 2 vs Cohort 3 vs Cohort 1EXT vs Cohort 2EXT vs Cohort 3EXT; The analysis compared the differences at Day 14 between aqueous gel (control) and vehicle gel (active Cohort 4 only) in abundance of Malassezia based on molecular diagnostic qPCR using a 2-sided Wilcoxon sign rank test, alpha = 0.05, with a null hypothesis of median difference equal to zero; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney); Mean Paired Change from Baseline = -483

2. Secondary Outcome: Proportion of Participants With Decrease in Signs and Symptoms of Tinea Versicolor for the DBI-002 DP-treated Lesion Compared to the Aqueous Gel Treated Lesion
Description: The secondary analysis will summarize the number of subjects with more improvement in individual signs and symptoms of TV between DBI-002 Drug Product (Active) and aqueous gel (Control) at Day 5 or Day 14 versus Baseline
Time Frame: 14 days of participation
Population: The proportion of subjects with a greater decrease in the scoring of individual signs and symptoms of TV for the DBI-002 Drug Product-treated lesion than the vehicle-treated or aqueous gel-treated lesion is be summarized descriptively for Days 5 and 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 1EXT | Cohort 2EXT | Cohort 3EXT
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 4 | 4
Participants
  Day 5 proportion of subjects with a greater decrease in the scoring of individual signs and symptoms | 2 | 2 | 2 | 2 | 1 | 2
  Day 14 proportion of subjects with a greater decrease in the scoring of individual signs and symptom | 3 | 3 | 3 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 14 (Visit 6) from the baseline Day 1 (Visit 1)
Description: AE is any untoward medical occurrence in a subject administered a pharmaceutical product, that doesn't necessarily have a causal relationship with the treatment.It can be any unfavorable & unintended sign(e.g., an abnormal laboratory finding), symptom/ disease temporally associated with use of the study drug, whether or not it's considered to be drug related.This includes any newly occurring event/previous condition that has increased in severity/frequency since the administration of study drug.
Groups:
- Cohort 1 Probiotic Gel; Cohort 1 Aqueous Gel; Cohort 1EXT Aqueous Gel; Cohort 1EXT Probiotic Gel: Low dose 10^6 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Cohort 2 Probiotic Gel; Cohort 2 Aqueous Gel; Cohort 2EXT Aqueous Gel; Cohort 2EXT Probiotic Gel: Medium dose 10^8 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Cohort 3 Aqueous Gel; Cohort 3 Probiotic Gel; Cohort 3EXT Aqueous Gel; Cohort 3EXT Probiotic Gel: High dose 10^10 CFUs /ml of DBI-002 probiotic vs. aqueous gel
  Single treatment dose OR Once-daily application for 5 consecutive days
- Cohort 4 Aqueous; Cohort 4 Probiotic: Vehicle gel vs. aqueous (CMC) gel Once-daily application for 5 consecutive days
Arm/Group | Cohort 1 Probiotic Gel | Cohort 1 Aqueous Gel | Cohort 2 Probiotic Gel | Cohort 2 Aqueous Gel | Cohort 3 Aqueous Gel | Cohort 3 Probiotic Gel | Cohort 1EXT Aqueous Gel | Cohort 1EXT Probiotic Gel | Cohort 2EXT Aqueous Gel | Cohort 2EXT Probiotic Gel | Cohort 3EXT Aqueous Gel | Cohort 3EXT Probiotic Gel | Cohort 4 Aqueous | Cohort 4 Probiotic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 1/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Probiotic Gel (N=6) | Cohort 1 Aqueous Gel (N=6) | Cohort 2 Probiotic Gel (N=6) | Cohort 2 Aqueous Gel (N=6) | Cohort 3 Aqueous Gel (N=6) | Cohort 3 Probiotic Gel (N=6) | Cohort 1EXT Aqueous Gel (N=4) | Cohort 1EXT Probiotic Gel (N=4) | Cohort 2EXT Aqueous Gel (N=4) | Cohort 2EXT Probiotic Gel (N=4) | Cohort 3EXT Aqueous Gel (N=4) | Cohort 3EXT Probiotic Gel (N=4) | Cohort 4 Aqueous (N=4) | Cohort 4 Probiotic (N=4)
Headache (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04937920/Prot_SAP_000.pdf